CLINICAL TRIAL: NCT02975297
Title: Exenatide Once Weekly for Smoking Cessation: A Randomized Clinical Trial
Brief Title: Exenatide Once Weekly for Smoking Cessation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Luba Yammine, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-17-0802; CCTS Research Scholar Award (Other: UTHealth)
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Smoking Cessation
Keywords: smoking; pre-diabetes; overweight; exenatide; Glucagon-like peptide-1 (GLP-1) agonists
MeSH Terms: conditions — Smoking Cessation; Smoking; Glucose Intolerance; Overweight | interventions — Exenatide; Tobacco Use Cessation Devices; Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exenatide plus NRT plus counseling (Experimental): Once weekly exenatide Injectable Product, Nicotine Replacement Therapy (NRT) Patch, smoking cessation counseling
  Interventions: Drug: Exenatide; Drug: NRT; Behavioral: Counseling
- Placebo plus NRT plus counseling (Placebo Comparator): Once weekly placebo, Nicotine Replacement Therapy (NRT) Patch, smoking cessation counseling
  Interventions: Drug: NRT; Behavioral: Counseling; Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Exenatide Injectable Product will be administered at a dose of 2 mg subcutaneously once a week for 6 weeks.
  Other Names: Bydureon
  Arms: Exenatide plus NRT plus counseling
Drug: NRT — Nicotine Patch (21mg) / 24 hours.
  Other Names: Nicotine patch
Behavioral: Counseling — Brief individual behavioral smoking cessation counseling.
  Other Names: Smoking cessation counseling
Drug: Placebo — Normal saline.
  Arms: Placebo plus NRT plus counseling

SUMMARY:
The purpose of this study is to identify a potential new treatment for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Be English-speaking volunteers who desire to quit smoking and are willing to make a quit attempt during the course of the study;
* Have smoked ≥10 cigarettes a day for at least one year and provide a breath carbon monoxide (CO) ≥10 ppm;
* Have a negative pregnancy test, if female of childbearing potential;
* Have HbA1C levels between 5.7 and 6.4% or BMI of or greater than 25 kg/square meters
* Not currently using any therapy for glycemic control (either injectable [i.e. insulin] or oral agents);
* Have vital signs as follows: resting pulse between 50 and 95 bpm, BP between 90-150 mmHg systolic and 45-95 mmHg diastolic;
* Have hematology and chemistry laboratory tests that are within reference limits (within 10% above or below), with the following exception: pancreatic tests (lipase and amylase) must be within normal limits;
* Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the principal investigator.

Exclusion Criteria:

* Meet criteria for the following psychiatric and/or substance use disorders as assessed by the Mini International Neuropsychiatric Interview (MINI): items C (current manic or hypomanic episode only), I (alcohol abuse - Alcohol Addendum-past 3 months only; current alcohol dependence), J (substance abuse -Substance Abuse Addendum - past 3 months only; current substance dependence), K (current psychotic disorder or current mood disorder with psychotic features).
* Individuals who meet criteria for non-exclusionary psychiatric disorders that are considered clinically unstable and/or unsuitable to participate as determined by the Principal Investigator and/or Study Physician.
* Individuals rated as moderate (9-16) to high (17 or greater) on suicidality as assessed by Module B of the MINI.
* Have personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2;
* Have type 1 diabetes mellitus;
* Have severe cardiovascular disease (history of myocardial infarction, life-threatening arrhythmia, or worsening angina pectoris);
* Have active temporomandibular joint disease;
* Have severe gastrointestinal disease (i.e. severe gastroparesis);
* Have previous history of pancreatitis or are at risk for pancreatitis;
* Have creatinine clearance (CrCl) < 30;
* Have any previous medically adverse reaction to study medications, nicotine, or menthol;
* Be pregnant or lactating or unwilling to provide a negative pregnancy test before study entry;
* Not using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide);
* Have any illness which in the opinion of the primary investigator would preclude safe and/or successful completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luba Yammine, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yammine L, Kosten TR, Cinciripini PM, Green CE, Meininger JC, Minnix JA, Newton TF. Exenatide once weekly for smoking cessation: study protocol for a randomized clinical trial. Medicine (Baltimore). 2018 Jan;97(2):e9567. doi: 10.1097/MD.0000000000009567. PMID 29480848
- [Derived] Yammine L, Green CE, Kosten TR, de Dios C, Suchting R, Lane SD, Verrico CD, Schmitz JM. Exenatide Adjunct to Nicotine Patch Facilitates Smoking Cessation and May Reduce Post-Cessation Weight Gain: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2021 Aug 29;23(10):1682-1690. doi: 10.1093/ntr/ntab066. PMID 33831213

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant in the exenatide arm did not receive exenatide, and 1 participant in the placebo arm did not receive placebo.
Period: Overall Study
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Started | 41 | 41
Completed | 34 | 35
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (9.1) | 51.2 (9.4) | 51.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 28 | 29 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 25 | 27 | 52
  White | 14 | 13 | 27
  Hispanic/Latino | 0 | 1 | 1
  Other | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 41 | 82
Marital Status [Count of Participants; unit: Participants]
  Never Married | 17 | 14 | 31
  Divorced/Separated | 17 | 20 | 37
  Married | 6 | 4 | 10
  Widowed | 1 | 3 | 4
Highest Level of Education [Count of Participants; unit: Participants]
  8th Grade or Less | 1 | 2 | 3
  High School | 27 | 24 | 51
  College Degree | 11 | 12 | 23
  Graduate Degree | 2 | 3 | 5
Household Income [Count of Participants; unit: Participants]
  <$19,999 | 23 | 26 | 49
  $20,000-39,999 | 12 | 10 | 22
  $40,000-59,999 | 2 | 2 | 4
  $60,000-79,999 | 4 | 0 | 4
  $80,000-99,999 | 0 | 1 | 1
  >$100,000 | 0 | 1 | 1
  Not reported | 0 | 1 | 1
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: Cigarettes Smoked per Day] | 18.5 (8.7) | 18.4 (9.3) | 18.4 (8.9)
Years of Regular Smoking [Mean (Standard Deviation); unit: years] | 27.4 (11) | 26.6 (12.7) | 27.0 (11.8)
Nicotine Dependence as Assessed by the Fagerstrom Test for Nicotine Dependence (FTND) [Mean (Standard Deviation); unit: score on a scale] — Total score ranges from 0-10. The higher the total Fagerström score, the more intense the physical dependence on nicotine.
  score on a scale | 6.3 (1.9) | 6 (2.5) | 6.2 (2.2)
Positive Affect as Assessed by the Positive and Negative Affect Schedule (PANAS) [Mean (Standard Deviation); unit: score on a scale] — Score ranges from 10-50, with a higher score representing higher levels of Positive Affect.
  score on a scale | 35.9 (10.1) | 32.5 (9.8) | 34.2 (10)
Negative Affect as Assessed by the Positive and Negative Affect Schedule (PANAS) [Mean (Standard Deviation); unit: score on a scale] — Score ranges from 10-50, with a higher score representing higher levels of Negative Affect.
  score on a scale | 18.6 (7.6) | 20.1 (8.0) | 19.3 (7.8)
Depressive Symptoms as Assessed by the Patient Health Questionnaire (PHQ-8) [Mean (Standard Deviation); unit: score on a scale] — Total score ranges from 0 to 24, with a higher score indicating greater depression.
  score on a scale | 8.3 (6.4) | 8.6 (5.9) | 8.5 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Self-Reported Abstinence and Who Were Biochemically Verified as Abstinent Via Expired CO Level of ≤ 5ppm
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 41 | 41
Participants | 19 | 11

2. Primary Outcome: Post-quit Craving as Assessed by the Questionnaire of Smoking Urges
Description: Questionnaire of Smoking Urges (QSU) is a 10-item scale (total score range = 10-70, a lower score indicates lower cravings for cigarettes) that evaluates the intention and desire to smoke and anticipation of relief from withdrawal-associated negative affect.
Time Frame: 6 weeks
Population: Data were not collected for 7 participants in the Exenatide plus NRT plus counseling arm and 6 participants in the Placebo plus NRT plus counseling arm. Overall Number of Participants Analyzed reflects participants who completed the study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 34 | 35
score on a scale | 17.2 (11.0) | 16.9 (9.75)

3. Primary Outcome: Withdrawal Symptoms as Assessed by the Wisconsin Smoking Withdrawal Scale
Description: The Wisconsin Smoking Withdrawal Scale is a 28-item questionnaire designed to assess different aspects of the smoking withdrawal syndrome. Participants rate each item on a Likert scale from zero (strongly disagree) to four (strongly agree). Total score ranges from 0 to 112, with a higher score indicating greater withdrawal.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 34 | 35
score on a scale | 40.5 (18.3) | 44.5 (18.0)

4. Primary Outcome: Cue-induced Craving for Cigarettes Following Virtual Reality Exposure as Assessed by the Questionnaire of Smoking Urges
Description: as for outcome 2
Time Frame: 1 week
Population: Virtual reality exposure was not done due to transfer of the study to a different site; therefore, data for this outcome measure were not collected.
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Cue-induced Craving for Cigarettes Following Virtual Reality Exposure as Assessed by the Questionnaire of Smoking Urges
Description: as for outcome 2
Time Frame: 3 weeks
Population: as for outcome 4
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Who Self-Reported Abstinence and Who Were Biochemically Verified as Abstinent Via Expired CO Level of ≤ 5ppm
Time Frame: 7 weeks (1 week after end of treatment)
Population: Data were not collected for 22 participants in the Exenatide plus NRT plus counseling arm and 30 participants in the Placebo plus NRT plus counseling arm. The Overall Number of Participants Analyzed reflects the number of participants who were abstinent [self-reported and verified by expired carbon monoxide (CO) levels (CO≤5 ppm)] at 6 weeks (end of treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 19 | 11
Participants | 15 | 7

7. Secondary Outcome: Number of Participants Who Self-Reported Abstinence and Who Were Biochemically Verified as Abstinent Via Expired CO Level of ≤ 5ppm
Time Frame: 10 weeks (4 weeks after end of treatment)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 19 | 11
Participants | 9 | 4

8. Secondary Outcome: Post-quit Craving as Assessed by the Questionnaire of Smoking Urges
Description: as for outcome 2
Time Frame: 7 weeks (1 week after end of treatment)
Population: Data were not collected for 25 participants in the Exenatide plus NRT plus counseling arm and 32 participants in the Placebo plus NRT plus counseling arm. The Overall Number of Participants Analyzed reflects those who completed the study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 16 | 9
score on a scale | 13.3 (7.86) | 14.2 (8.47)

9. Secondary Outcome: Post-quit Craving as Assessed by the Questionnaire of Smoking Urges
Description: as for outcome 2
Time Frame: 10 weeks (4 weeks after end of treatment)
Population: Data were not collected for 30 participants in the Exenatide plus NRT plus counseling arm and 37 participants in the Placebo plus NRT plus counseling arm. The Overall Number of Participants Analyzed reflects those who completed the study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
Number analyzed (Participants) | 11 | 4
score on a scale | 11.5 (5.13) | 11.2 (2.5)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Exenatide Plus NRT Plus Counseling | Placebo Plus NRT Plus Counseling
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 4/41 | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide Plus NRT Plus Counseling (N=41) | Placebo Plus NRT Plus Counseling (N=41)
Injection site nodule (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Pruritus at the site of nicotine patch application (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT02975297/Prot_SAP_000.pdf